CLINICAL TRIAL: NCT01324700
Title: Antidepressant Treatment at an Inner City Asthma Clinic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 072010-235; R18HL092862 (NIH)
Record Dates: First submitted 2010-10-19; First posted 2011-03-29 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Depression; Asthma
MeSH Terms: conditions — Depression; Asthma | interventions — Escitalopram; Selective Serotonin Reuptake Inhibitors; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High severity group: Escitalopram (Active Comparator): Participants with Baseline score of 20 or above on the 17-item Hamilton Rating Scale for Depression (HRSD) AND 3 or more courses of oral corticosteroids in the past 12 months were stratified into high severity group. Then these participants were further stratified into escitalopram group.
  Interventions: Drug: High severity group: Escitalopram
- Low severity group: Escitalopram (Active Comparator): Participants with Baseline HRSD score of less than 20 AND fewer than 3 courses of oral corticosteroids in the past 12 months were stratified into low severity group. Then these participants were further stratified into escitalopram group.
  Interventions: Drug: Low severity group: Escitalopram
- High severity group: Placebo (Placebo Comparator): Participants with Baseline score of 20 or above on the 17-item Hamilton Rating Scale for Depression (HRSD) AND 3 or more courses of oral corticosteroids in the past 12 months were stratified into high severity group. Then these participants were further stratified into placebo group.
  Interventions: Drug: High severity group: Placebo
- Low severity group: Placebo (Placebo Comparator): Participants with Baseline HRSD score of less than 20 AND fewer than 3 courses of oral corticosteroids in the past 12 months were stratified into low severity group. Then these participants were further stratified into placebo group.
  Interventions: Drug: Low severity group: Placebo

INTERVENTIONS:
Drug: High severity group: Escitalopram — Participants within high severity group were stratified to receive escitalopram.
  Other Names: Lexapro, Selective serotonin reuptake inhibitor (SSRI)
  Arms: High severity group: Escitalopram
Drug: High severity group: Placebo — Participants within high severity group were stratified to receive placebo (inactive ingredient matching the active medication in appearance).
  Other Names: Sugar pill
  Arms: High severity group: Placebo
Drug: Low severity group: Escitalopram — Participants within low severity group were stratified to receive escitalopram.
  Other Names: Lexapro, Selective serotonin reuptake inhibitor (SSRI)
  Arms: Low severity group: Escitalopram
Drug: Low severity group: Placebo — Participants within low severity group were stratified to receive placebo (inactive ingredient matching the active medication in appearance).
  Other Names: Sugar pill
  Arms: Low severity group: Placebo

SUMMARY:
Asthma is common with an increasing prevalence and mortality especially in low-income and minority populations. The course of asthma appears to be influenced by mood and emotions. It has been reported that there is a high prevalence of depression or depressive symptoms in both children and adults with asthma. Despite data on the frequency of depression in asthma and its adverse consequences, it is generally not recognized or treated. Brown et al. conducted a randomized, double-blind, placebo-controlled trial of citalopram in 90 outpatients with asthma and MDD. Citalopram therapy was associated with lower depression scores, numerically greater rates of remission of depressive symptoms, and less oral corticosteroid use than placebo. The investigators proposed study is different. The investigators observed a modest difference between antidepressant and placebo in the prior trial. However, in a subgroup with more severe asthma (based on frequent corticosteroid use) and more severe depression (based on higher depressive symptoms scores) the investigators saw a much larger effect size. Standard of care for severe asthma is aggressive asthma treatment. The investigators study does not require any changes in the patient's asthma treatment. No guidelines are currently available on the treatment of depression in asthma patients. Standard care for depression would be antidepressants.

DETAILED DESCRIPTION:
A 12-week, randomized, double-blind, parallel-group, placebo-controlled acute phase trial of escitalopram is proposed in 222 persons with asthma and Major Depressive Disorder (MDD). This sample will consist of 80 stratified into the High severity group which will consist of a baseline score > or = 20 on the 17-item Hamilton Rating Scale for Depression (HRSD) and > or = 3 courses of oral corticosteroids in the past 12 months. A separate group stratified into the Low severity group of 142 with MDD and asthma but HRSD-17 scores of < 20 and < 3 courses of oral corticosteroids in the past 12 months. A 16 week continuation phase is also proposed for depression responders at week 12. The participants will be recruited at the Parkland Hospital Health System (PHHS) Asthma and Allergy Clinics and Aston Clinic using the Self-Report Screening Tool for Depression (2-SRSD), a brief depression questionnaire, as part of routine clinical practice. Potential participants will be given an appointment scheduled at the PI's office to complete baseline assessment at which time written informed consent will be obtained before any study-specific assessments are completed. At the baseline appointment, the RA will administer the Structured Clinical Interview for DSM-IV (SCID) at baseline to establish a current diagnosis of MDD. Participants meeting all inclusion criteria will then be administered the IDS-SR30, the SF-36, the Asthma Control Questionnaire (ACQ), Mini Asthma Quality of Life Questionnaire (Mini AQLQ), the Cumulative Illness Rating Scale (CIRS), the PRD-III Somatic Symptom Scale (PRD-III) for side effects, a blood draw for routine laboratory analyses, and forced expiratory volume in 1-second percentage of normal (FEV1%) will be assessed using a portable spirometer. Self-reported asthma-related emergency room visits and hospitalizations will be quantified for the past 12 months.

Participants will receive a clinical psychiatric evaluation by one of the investigators to confirm the diagnosis and that the participant meets entry criteria. Steroid inhaler dose monitoring using the counter already included by the manufacturer will begin at this time. After the participant is determined to qualify, the steroid inhaler counter will be used to assess baseline adherence. Participants will be randomized and receive either escitalopram or a placebo identical in appearance. Each participant will then be given a 14-day supply of active medication (escitalopram 10 mg) or placebo and asked to return for a follow-up appointment in two weeks. Each participant will be given a phone number to reach the Principle Investigator (PI) and Research Assistant (RA) 24 hours a day. The RA will obtain written consent to inform the physician treating their asthma of their participation in the study. Each participant will then return for follow-up appointments twice per month at which time they will repeat the outcome measures according to the schedule given below. Pill counts will be conducted, MEMS caps analyzed and a list of current medications and doses will be obtained at each visit. Participants will be evaluated by both the RA and PI at each follow-up appointment. Participants who have not shown evidence of adequate response (< 30% decrease in HRSD) to the antidepressant at week 4, and who do not have side effects, will have the dose increased to two tablets (20 mg of active medication or placebo). At week 12, responders (HRSD reduction ≥50% from baseline) will continue on blinded treatment with assessments every 4 weeks for an additional 16 weeks (continuation phase). Nonresponders will be removed from the study and given standard treatment by an unblinded psychiatrist (Dr. Nakamura) until referral can be made for further treatment. Continuation phase will begin at the final week 12 assessment for responders. They will be given a 4-week supply of medication at the dose they are taking at week 12, and instructions to call if they experience a worsening in symptoms (e.g., decrease in sleep, suicidal thoughts) between the 4-week appointments, and an appointment with a study physician will be arranged. The HRSD will be assessed at any interim appointments and the participant discontinued if they meet discontinuation criteria. Treatment referral will be arranged as in the acute phase study. At completion of 28 weeks, they will be referred for further treatment as appropriate, with their PCP, the Parkland Psychiatry Clinic, a private psychiatrist, a UT Southwestern Medical Center, or the county Mental Health Mental Retardation (MHMR) system. Parking/bus tokens will be provided. A final visit for safety, to assess follow-up adherence and collect asthma and depression outcome data will be arranged 4 weeks after the last appointment (e.g., discontinuation at end of acute phase, end of continuation phase, or if discontinued early for any reason).

The assessment schedule is designed to approximate good clinical practice for depression and, thus, may be somewhat less intensive than in some antidepressant trials. The following assessment instruments will be used in this investigation. A two-item, self-report screening tool for depression (2-SRSD) taken from the Primary Care Evaluation of Mental Disorders Procedure (PRIME-MD) screening interview will be used to detect suspected cases of depression among asthma clinic patients. The specificity of the 2-SRSD in this population was 57%. Thus, we expect to identify almost all true positives, with a substantial number of false positives. A positive answer to either 1) "During the past month, have you often been bothered by feeling down, depressed, or hopeless?" or 2) "During the past month, have you often been bothered by little interest or pleasure in doing things?" will be considered a possible case of depression and qualify for further assessment. MDD is defined as at least five of nine symptoms that must include depressed mood or loss of interest and can also include psychomotor changes, appetite changes or weight loss, sleep changes, decreased concentration, guilt, decreased energy levels (lassitude), and suicidal ideation. The symptoms must occur at the same time and last for at least 2 weeks and be associated with a change in functioning. The symptoms must not be the direct physiologic effect of a drug or medical illness (e.g., hypothyroidism) or bereavement. MDD is diagnosed using a structured clinical interview that addresses each symptom and uses information from the patient, family, physicians, and medical records to establish the diagnosis.

The clinician version of the structured Clinical Interview for DSM-IV (SCID) is a brief structured interview for major Axis I disorders in DSM-IV including major depressive disorder, dysthymic disorder, bipolar disorders, psychotic disorders, anxiety disorders, eating disorders, and alcohol and substance abuse/dependence. The Hamilton Rating Scale for Depression (HRSD, 17-item version) is an observer-rated measure of depressive symptomatology. The HRSD will be administered at every visit. The Inventory of Depressive Symptomatology-Self-report (IDS-SR30) is a 30-item self-report scale that assesses depressive symptom severity. The IDS-SR30 will be administered at every visit. The Hamilton Rating Scale for Anxiety (HRSA) is a 14-item observer rating scale that assesses the degree and pathology associated with anxiety such as anxious mood, tension, fear, and insomnia. The HRSA will be administered at every visit. Asthma symptoms will be assessed at every visit using the Asthma Control Questionnaire (ACQ). Pulmonary function will also be assessed at every visit by spirometry, using equipment meeting the standards of the ATS, and calibrated according to the manufacturer's recommendations. Spirometry will be performed according to ATS guidelines, as the best of three acceptable efforts. Spirometry will be measured before, and 10 minutes after, two puffs of albuterol are administered via metered dose inhaler. Bronchodilator response is calculated as [(post FEV1 - pre FEV1)/pre FEV1], and converted to a percent improvement.

The Psychobiology of Recovery in Depression-III Somatic Symptom Scale (PRD-III) is a 24 item, side effects scale developed for a longitudinal depression study. The PRD-III covers a wide range of common medication side effects and can be quickly and easily administered by a clinician. The PRD-III will be administered at every visit. Asthma-related quality of life will be assessed with the Mini-AQLQ, a 15 item, self-administered scale measuring functional impairments troublesome to adult asthma patients. Mini-AQLQ showed good responsiveness, reliability, and construct validity compared to the longer 32 item version. Both versions of the Mini-AQLQ correlate well with SF 36 mental and physical subscales and ACQ scores (asthma symptoms), but not with spirometry or beta-agonist use. The Mini-AQLQ will be administered at baseline, week 4, week 8, week 12, and at exit or if continued, week 28. General functioning will be assessed with the 36-Item Short Form Health Survey (SF-36), a self-reported tool used to assess physical and mental functioning. The scale consists of summary measures of physical and mental health that can be further divided into scales for physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores above the normative score of 50±10 indicate better than average functioning while scores below 50 suggest below normal functioning. The SF-36 will be administered at baseline, week 4, week 8, week 12, and at exit or if continued, week 28.

Medical illness burden will be assessed at baseline and at exit with the Cumulative Illness Rating Scale (CIRS), a valid and widely used 13-item, 0-4, clinician-rated scale that assesses medical impairment related to major organ systems. Medical history and review of systems is used for the rating. The scale will be rated by a study physician. The scale has been used in other recent antidepressant trials to assess medical illness burden. The Perceived Stress Scale (PSS-10) is a 10-item, 0-4 self-report scale that assesses stressful feelings and thoughts in the past month. The PSS-10 has adequate reliability and validity and is a better predictor of some outcomes (e.g. depressive and physical symptoms, utilization of health services, social anxiety) than were life-event scores. The PSS-10 appears to provide a general appraisal of life stress. The PSS-10 will be administered at baseline, week 4, week 8, week 12, and at exit or if continued, week 28.

Specific Primary and Secondary Outcome Measures associated with primary and secondary aims include:

Primary Aim:

1. Escitalopram treatment will be associated with greater improvement in asthma symptoms, using ACQ measure, than placebo in outpatients with asthma and MDD.

Secondary Aim:

1. Escitalopram treatment will be associated with greater depressive symptom remission rates, using HRSD, than placebo in outpatients with asthma and MDD.

ELIGIBILITY:
Inclusion Criteria:

* Acute phase:

  * Physician diagnosis of asthma and currently receiving asthma treatment, Current diagnosis of MDD confirmed by the SCID and clinical assessment by a psychiatrist
  * Baseline HRSD ≥ 15
  * Baseline ACQ score of ≥ 1
  * Ages 18-70 years to include the range of ages typically treated at our referral sources
  * No changes in asthma medications, oral corticosteroid use, or treatment for respiratory tract infections in the past 2 weeks
  * Both male and female
  * English- or Spanish-speaking
* Continuation phase:

  * Completed week 12 assessment of acute treatment phase
  * Acute phase responders (defined as a baseline to week 12 reduction in the HRSD score of 50% or greater)

Exclusion Criteria:

* Acute phase:

  * Current substance and alcohol abuse/dependence
  * Current daily tobacco use
  * Severe or life threatening medical illness that would make completion of study unlikely (e.g. myocardial infarction)
  * MDD with psychotic features (delusions, hallucinations, disorganized thought processes, etc), bipolar disorder, schizophrenia, schizoaffective disorder, or substance-induced mood disorder and mood disorders secondary to a general medical condition
  * Vulnerable populations including mentally retarded persons or those with other severe cognitive impairment, prison or jail inmates, pregnant or nursing women or women of childbearing age who will not use UTSW IRB-approved methods of birth control or abstinence during the study
  * Initiation on other psychotropic medications within the past 2 weeks
  * High risk for suicide defined as > 1 past attempts or current suicidal ideation with plan and intent or HRSD suicide question score of ≥ 2
  * Use of antidepressants at therapeutic doses for depression within 1 week of study entry. Potential participants taking antidepressants (other than escitalopram) for depression may be enrolled following 1 week washout if they currently meet depression entry criteria and have been taking the medication for at least 4 weeks at a therapeutic dose (non-responder)
  * Patients currently taking but not responding to escitalopram (current study drug). At week 8, if HRSD is < 25% decrease from HRSD baseline score, clinician may consider discontinuation since response by week 12 in these patients is unlikely
* Continuation phase:

  * Development of exclusion criteria for acute phase (i.e., current suicidal ideation with plan and intent)
  * HRSD score > 50% of baseline score (no longer meets criteria as a responder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System (Asthma, Allergy, & Arthritis Clinics), Dallas, Texas, United States

REFERENCES:
- [Derived] Agarwal CD, Palka JM, Gajewski AJ, Khan DA, Brown ES. The efficacy of citalopram or escitalopram in patients with asthma and major depressive disorder. Ann Allergy Asthma Immunol. 2024 Mar;132(3):374-382. doi: 10.1016/j.anai.2023.11.004. Epub 2023 Nov 11. PMID 37952772

RESULTS

PARTICIPANT FLOW:
Groups:
- High Severity: Escitalopram: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). To be assigned to the high severity group, participants had to have at least 3 steroid bursts in the past 12 months AND Hamilton Rating Scale for Depression (HRSD) score of at least 20. Participants received escitalopram (or identical placebo) at the dose of 10 mg/day with follow-up visits every 2 weeks for 12 total weeks. Participants who had not shown a decrease in HRSD score of at least 30% by week 4, had their dosage of escitalopram increased to 20 mg/day (or equivalent placebo).
- High Severity: Placebo: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). To be assigned to the high severity group, participants had to have at least 3 steroid bursts in the past 12 months AND Hamilton Rating Scale for Depression (HRSD) score of at least 20. Participants received placebo (identical in appearance to the active medication) with follow-up visits every 2 weeks for 12 total weeks.
- Low Severity: Escitalopram: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). To be assigned to the low severity group, participants had to have fewer than 3 steroid bursts in the past 12 months OR Hamilton Rating Scale for Depression (HRSD) score of less than 20 (or both). Participants received escitalopram (or identical placebo) at the dose of 10 mg/day with follow-up visits every 2 weeks for 12 total weeks. Participants who had not shown a decrease in HRSD score of at least 30% by week 4, had their dosage of escitalopram increased to 20 mg/day (or equivalent placebo).
- Low Severity: Placebo: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). To be assigned to the low severity group, participants had to have fewer than 3 steroid bursts in the past 12 months OR Hamilton Rating Scale for Depression (HRSD) score of less than 20. Participants received placebo (identical in appearance to the active medication) with follow-up visits every 2 weeks for 12 total weeks.
Period: Overall Study
Arm/Group | High Severity: Escitalopram | High Severity: Placebo | Low Severity: Escitalopram | Low Severity: Placebo
Started | 22 | 20 | 49 | 48
Completed | 13 | 16 | 33 | 37
Not Completed | 9 | 4 | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- High Severity: Escitalopram: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). Participants in the "high severity-escitalopram" group had at least 3 steroid bursts in the past 12 months AND Hamilton Rating Scale for Depression (HRSD) score of at least 20. Participants received oral escitalopram at the dose of 10 mg/day with follow-up visits every 2 weeks for 12 total weeks. Participants who had not shown a decrease in HRSD score of at least 30% by week 4, had their dosage of escitalopram increased to 20 mg/day.
- High Severity: Placebo: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). Participants in the "high severity-placebo" group had at least 3 steroid bursts in the past 12 months AND Hamilton Rating Scale for Depression (HRSD) score of at least 20. Participants received oral placebo (identical in appearance to the active medication) every 2 weeks for 12 total weeks.
- Low Severity: Escitalopram: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). Participants in the "low severity-escitalopram" group had at least 3 steroid bursts in the past 12 months OR Hamilton Rating Scale for Depression (HRSD) score of at least 20. Participants received oral escitalopram at the dose of 10 mg/day with follow-up visits every 2 weeks for 12 total weeks. Participants who had not shown a decrease in HRSD score of at least 30% by week 4, had their dosage of escitalopram increased to 20 mg/day.
- Low Severity: Placebo: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description). Participants in the "low severity-placebo" group had at least 3 steroid bursts in the past 12 months OR Hamilton Rating Scale for Depression (HRSD) score of at least 20. Participants received oral placebo (identical in appearance to the active medication) every 2 weeks for 12 total weeks.
- Total: Total of all reporting groups
Arm/Group | High Severity: Escitalopram | High Severity: Placebo | Low Severity: Escitalopram | Low Severity: Placebo | Total
Number analyzed (Participants) | 22 | 20 | 49 | 48 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.50 (12.34) | 45.85 (11.17) | 44.51 (12.08) | 43.92 (11.60) | 44.18 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 39 | 31 | 100
  Male | 5 | 7 | 10 | 17 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 11 | 29 | 28 | 83
  White | 6 | 9 | 19 | 19 | 53
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (ACQ)
Description: The ACQ has 7 questions (the top scoring 5 symptoms, FEV1% pred. and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). Clinic staff score the FEV1% predicted on a 7-point scale. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Severity: Escitalopram; High Severity: Placebo; Low Severity: Escitalopram; Low Severity: Placebo: Participants were stratified into high vs. low severity groups, and then further stratified into escitalopram or placebo groups (see study arm/intervention description).
Arm/Group | High Severity: Escitalopram | High Severity: Placebo | Low Severity: Escitalopram | Low Severity: Placebo
Number analyzed (Participants) | 13 | 16 | 33 | 37
units on a scale | 1.15 (0.48) | 1.63 (0.89) | 1.39 (0.20) | 1.23 (0.92)

2. Secondary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: The patient is rated by a clinician on 17 items that measure depressive symptom severity. The total score is calculated by summing the responses across all items. Lower scores (closer to 0) indicate the absence of depressive symptoms, while higher scores indicate the presence of depressive symptoms. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2 (0 = not present; 2 = severe). The scale range of scores is 0-52.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Severity: Escitalopram | High Severity: Placebo | Low Severity: Escitalopram | Low Severity: Placebo
Number analyzed (Participants) | 13 | 16 | 33 | 37
units on a scale | 10.08 (6.54) | 14.38 (8.69) | 10.39 (8.07) | 9.31 (6.00)

ADVERSE EVENTS:
Arm/Group | High Severity: Escitalopram | High Severity: Placebo | Low Severity: Escitalopram | Low Severity: Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 1/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 2/22 | 8/20 | 5/49 | 7/48
Other Adverse Events (participants affected / at risk) | 4/22 | 1/20 | 5/49 | 9/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Severity: Escitalopram (N=22) | High Severity: Placebo (N=20) | Low Severity: Escitalopram (N=49) | Low Severity: Placebo (N=48)
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Congestive heart failure (Cardiac disorders) | 0 | 2 | 0 | 0
Dehydration (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 3
Chest pain (Cardiac disorders) | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Hypertensive cardiovascular disease (Cardiac disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Fall (Social circumstances) | 0 | 0 | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Severity: Escitalopram (N=22) | High Severity: Placebo (N=20) | Low Severity: Escitalopram (N=49) | Low Severity: Placebo (N=48)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 3
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Precancerous labial cells (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Kidney infection (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Yeast infection (Infections and infestations) | 0 | 0 | 1 | 0
Acid reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fainting (Vascular disorders) | 0 | 0 | 0 | 1
Dizziness (Vascular disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No